CLINICAL TRIAL: NCT02921919
Title: A SINGLE-ARM, OPEN-LABEL, MULTICENTER, EXTENDED TREATMENT, SAFETY STUDY IN PATIENTS TREATED WITH TALAZOPARIB
Brief Title: Open-Label Extension and Safety Study of Talazoparib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-13; C3441010 (Other: Alias Study Number); 2016-001972-31 (EudraCT Number)
Record Dates: First submitted 2016-09-22; First posted 2016-10-03 (Estimated); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — talazoparib

ARMS (1):
- Talazoparib (Experimental)
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Maximum starting dose: 1mg/day or last tolerated dose in the originating protocol
  Other Names: MDV3800

SUMMARY:
This is a single-arm, open-label, extended treatment, safety study in patients treated with talazoparib in qualifying studies.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Female patients of childbearing potential must have a negative pregnancy test before the first dose of talazoparib and must agree to use a highly effective birth control method from the time of the first dose of talazoparib through 45 days after the last dose.
* Male patients must use a condom when having sex with a pregnant woman or with a woman of childbearing potential from the time of the first dose of talazoparib through 105 days after the last dose. Contraception should be considered for a nonpregnant female partner of childbearing potential.
* Female patients may not be breastfeeding at the first dose of talazoparib and must not breastfeed during study participation through 45 days after the last dose of talazoparib.

Exclusion Criteria:

* Permanently discontinued from any Medivation sponsored study with talazoparib alone or in combination with another agent.
* Received an antineoplastic therapy or investigational agent after treatment with talazoparib in the originating protocol.
* Has a clinically significant cardiovascular, dermatologic, endocrine, gastrointestinal, hematologic, infectious, metabolic, neurologic, psychologic, or pulmonary disorder or any other condition, including excessive alcohol or drug abuse, or secondary malignancy, that may interfere with study participation in the opinion of the investigator.
* Diagnosis of myelodysplastic syndrome (MDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (24):
  - UCLA Hematology/Oncology - Alhambra, Alhambra, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - UCLA Hematology/Oncology - Burbank, Burbank, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Pharm.D., Los Angeles, California
  - (IRB# 16-001189) Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology - Pasadena, Pasadena, California
  - UCLA Hematology/Oncology - Porter Ranch, Porter Ranch, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Torrance Oncology, Torrance, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - Orlando Health, Inc., Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - IU Health Bloomington Hospital, Bloomington, Indiana
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Senvices, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Clinic, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Institut Paoli-Calmettes, Marseille, France
- Frauenklinik des Universitaetsklinikums Erlangen, Erlangen, Germany
- Hungary (2):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Onkologiai Osztaly, Budapest
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati-Onkologiai Osztaly es Klinikai Farmakologiai Osztaly, Budapest
- Arensia Exploratory Medicine, Institutia Medico-Sanitara Publica Institutul Oncologic, Chisinau, Moldova
- Szpital Lux Med, Warsaw, Poland
- Russia (2):
  - FSBEI HE " First Moscow State Medical University n.a. I.M. Sechenov" of the MoH of the RF, Moscow
  - Medical Technologies LLC, Saint Petersburg
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MDV3800-13

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who received talazoparib as a single agent or in combination with another agent in following qualifying studies: PRP-001(NCT01286987), MDV3800-01(NCT02997163), MDV3800-02(NCT02997176), MDV3800-03(NCT03070548), MDV3800-04(NCT03077607), MDV3800-14(NCT03042910) continued therapy with talazoparib as single agent in this extended treatment study.
Pre-assignment Details: A total of 120 participants were enrolled in the study of which 118 participants received the study treatment and 2 participants did not receive any study treatment as they were withdrawn before treatment initiation. Hence those 2 participants were not reported under any reporting arms.
Groups:
- Initial Dose Talazoparib: < 1 mg/Day: Participants were administered talazoparib capsules at an initial dose (i.e. the last tolerated dose in the originating study) of less than (<) 1 milligram (mg) orally once daily. Participants received talazoparib till the investigator considered treatment to be providing clinical benefit or until other study discontinuation criteria were met. Participants were followed-up for safety until 30 days after the last dose of talazoparib (i.e., permanent discontinuation) or before initiation of a new antineoplastic therapy, whichever occurred first.
- Initial Dose Talazoparib: 1 mg/Day: Participants were administered talazoparib capsules at an initial dose (i.e. the last tolerated dose in the originating study) of 1 mg orally once daily. Participants received talazoparib till the investigator considered treatment to be providing clinical benefit or until other study discontinuation criteria were met. Participants were followed-up for safety until 30 days after the last dose of talazoparib (i.e., permanent discontinuation) or before initiation of a new antineoplastic therapy, whichever occurred first.
Period: Overall Study
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Started | 66 | 52
Treated | 66 | 52
Completed | 0 | 0
Not Completed | 66 | 52
Not completed — Other | 5 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Disease Progression | 47 | 38
Not completed — Physician Decision | 3 | 2
Not completed — Adverse Event | 6 | 4

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included the participants who received any amount of talazoparib in this study.
Groups:
- Initial Dose Talazoparib: < 1 mg/Day: Participants were administered talazoparib capsules at an initial dose (i.e. the last tolerated dose in the originating study) of < 1 mg orally once daily. Participants received talazoparib till the investigator considered treatment to be providing clinical benefit or until other study discontinuation criteria were met. Participants were followed-up for safety until 30 days after the last dose of talazoparib (i.e., permanent discontinuation) or before initiation of a new antineoplastic therapy, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day | Total
Number analyzed (Participants) | 66 | 52 | 118
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 10 | 9 | 19
  50 to <65 years | 30 | 17 | 47
  >= 65 years | 25 | 25 | 50
  Missing | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 83
  Male | 20 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 56 | 45 | 101
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 59 | 48 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (SAEs), Treatment Emergent Treatment Related AEs and Treatment Emergent Treatment Related SAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a study drug without regard to possibility of a causal relationship. SAE was any untoward medical occurrence that at any dose resulted in death; inpatient hospitalization or prolongation of existing hospitalization; was life-threatening (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect or was considered as an important medical event. TEAEs were AEs that occurred on or after the administration of first dose of study drug through approximately 30 days after the last dose. AE included both SAEs and all non-SAEs. Treatment-related TEAEs were defined as any TEAE with at least a possible relationship to the study drug as assessed by the investigator or that was missing the assessment of causal relationship whose relationship to the study drug could not be ruled out.
Time Frame: From start of study treatment up to 30 days after last dose of study treatment or before initiation of a new antineoplastic therapy, whichever occurred first (approximately maximum for 4.6 years)
Population: Safety population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 66 | 52
Participants
  TEAE | 63 | 47
  SAE | 27 | 18
  Treatment-related TEAEs | 45 | 31
  Treatment-related SAEs | 6 | 3

2. Primary Outcome: Number of Participants With Grade 3 or 4 TEAEs Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4
Description: An AE was any untoward medical occurrence in a participant administered a study drug without regard to possibility of a causal relationship. TEAEs were AEs that occurred on or after the administration of first dose of study drug through approximately 30 days after the last dose. Severity was graded using NCI-CTCAE version 4 where, Grade 1: mild AE; Grade 2: moderate AE; Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated; Grade 5: death related to AE. Number of participants with Grade 3 or 4 TEAEs were reported.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 66 | 52
Participants | 38 | 32

3. Primary Outcome: Number of Participants With TEAEs Leading to Dose Reduction, Permanent Study Drug Discontinuation and Death
Description: An AE was any untoward medical occurrence in a participant administered a study drug without regard to possibility of a causal relationship. TEAEs were AEs that occurred on or after the administration of first dose of study drug through approximately 30 days after the last dose. Number of participants with TEAEs leading to dose reduction, permanent study drug discontinuation and death were reported.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 66 | 52
Participants
  TEAE leading to dose reduction | 6 | 7
  TEAE leading to permanent study drug discontinuation | 5 | 4
  TEAE leading to death | 7 | 7

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities: Liver Function Tests
Description: The following liver parameters were analyzed: aspartate transaminase (AST), alanine aminotransferase (ALT), total bilirubin (TBL) and alkaline phosphatase (ALP). The criteria for clinically significant abnormalities for liver parameters included AST or ALT greater than or equal to (>=) 3 times upper limit of normal (ULN); ALT or AST greater than (>) 5 times ULN; ALT or AST > 10 times ULN; ALT or AST > 20 times ULN; total TBL >2 times ULN; ALT or AST >= 3 times ULN and TBL > 2 times ULN and ALT or AST >= 3 times ULN and TBL > 2 times ULN and ALP < 2 times ULN.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any amount of talazoparib. Here, "overall number of participants analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 61 | 50
Participants
  ALT or AST >= 3*ULN | 5 | 2
  ALT or AST > 5*ULN | 0 | 0
  ALT or AST > 10*ULN | 0 | 0
  ALT or AST > 20*ULN | 0 | 0
  TBL > 2*ULN | 4 | 0
  ALT or AST >= 3*ULN and TBL > 2*ULN (any visit date) | 2 | 0
  ALT or AST >= 3*ULN and TBL > 2*ULN and ALP < 2*ULN (any visit date) | 0 | 0

5. Primary Outcome: Number of Participants With NCI-CTCAE Grade 3/4 Postbaseline Laboratory Toxicities: Hematology Parameters
Description: The following hematology parameters were analyzed: hemoglobin, leukocytes, lymphocytes, neutrophils and platelets. Laboratory toxicities were graded using NCI-CTCAE version 4 where, grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (potentially life threatening) and grade 5 (death) for each parameter. Number of participants with Grade 3 and 4 toxicities were reported. Low indicates values lower than the normal range.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 66 | 52
Participants
  Hemoglobin (low): Grade 3 | 7 | 16
  Hemoglobin (low): Grade 4 | 0 | 0
  Leukocytes (low): Grade 3 | 5 | 2
  Leukocytes (low): Grade 4 | 0 | 0
  Lymphocytes (low): Grade 3 | 11 | 8
  Lymphocytes (low): Grade 4 | 1 | 1
  Neutrophils (low): Grade 3 | 9 | 4
  Neutrophils (low): Grade 4 | 1 | 0
  Platelets (low): Grade 3 | 4 | 4
  Platelets (low): Grade 4 | 1 | 1

6. Primary Outcome: Number of Participants With NCI-CTCAE Grade 3/4 Postbaseline Laboratory Toxicities: Chemistry Parameters
Description: The following chemistry parameters were analyzed: alkaline phosphatase, bilirubin and creatinine. Laboratory toxicities were graded using NCI-CTCAE version 4 where, grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (potentially life threatening) and grade 5 (death) for each parameter. Number of participants with Grade 3 or 4 toxicities were reported. High indicates values higher than the normal range.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 66 | 52
Participants
  Alkaline Phosphatase (high): Grade 3 | 5 | 1
  Alkaline Phosphatase (high): Grade 4 | 1 | 0
  Bilirubin (high): Grade 3 | 3 | 0
  Bilirubin (high): Grade 4 | 1 | 0
  Creatinine (high): Grade 3 | 1 | 0
  Creatinine (high): Grade 4 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs and Weight
Description: Criteria for clinically significant changes in vital signs included a) Systolic blood pressure (SBP): 1) absolute results >180 millimeter of mercury (mmHg) and increase from baseline >=40 mmHg, 2) absolute results <90 mmHg and decrease from baseline >30 mmHg; b) Diastolic blood pressure (DBP): 1) absolute results >110 mmHg and increase from baseline >=30 mmHg , 2) absolute results <50 mmHg and decrease from baseline >20 mmHg , 3) increase from baseline >=20 mmHg; c) Heart rate: 1) absolute results >120 beats per minute (bpm) and increase from baseline >30 bpm, 2) absolute results <50 bpm and >20 bpm decrease from baseline; d) Temperature: <=34.5 or >=38 degree Celsius. Criteria for clinically significant changes in weight: >10 percent (%) decrease from baseline.
Time Frame: as for outcome 1
Population: Safety population included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
Number analyzed (Participants) | 66 | 52
Participants
  SBP: absolute results >180 mmHg and increase from baseline >=40 mmHg | 1 | 0
  SBP: absolute results <90 mmHg and decrease from baseline >30 mmHg | 1 | 0
  DBP: absolute results >110 mmHg and increase from baseline >=30 mmHg | 0 | 0
  DBP: absolute results <50 mmHg and decrease from baseline >20 mmHg | 0 | 0
  DBP: increase from baseline >=20 mmHg | 6 | 5
  Heart rate: absolute results >120 bpm and increase from baseline >30 bpm | 2 | 0
  Heart rate: absolute results <50 bpm and decrease from baseline >20 bpm | 0 | 0
  Temperature: <=34.5 or >=38 degree Celsius | 0 | 0
  Weight: >10% decrease from baseline | 7 | 2

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after last dose of study treatment or before initiation of a new antineoplastic therapy, whichever occurred first (approximately maximum for 4.6 years)
Description: An AE term may be reported as both a serious and non-serious AE, but are distinct events. An AE may be serious for 1 participant and non-serious for another participant, or a participant may have experienced both a serious and non-serious episode of the same event. Safety population included all participants who received any amount of talazoparib.
Arm/Group | Initial Dose Talazoparib: < 1 mg/Day | Initial Dose Talazoparib: 1 mg/Day
All-Cause Mortality (participants affected / at risk) | 7/66 | 8/52
Serious Adverse Events (participants affected / at risk) | 27/66 | 18/52
Other Adverse Events (participants affected / at risk) | 54/66 | 46/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose Talazoparib: < 1 mg/Day (N=66) | Initial Dose Talazoparib: 1 mg/Day (N=52)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Disease Progression (General disorders) | 4 | 0
Gait Disturbance (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Endocarditis Bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Streptococcal Sepsis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Failure To Thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Pericardial Effusion Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Cauda Equina Syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose Talazoparib: < 1 mg/Day (N=66) | Initial Dose Talazoparib: 1 mg/Day (N=52)
Anaemia (Blood and lymphatic system disorders) | 19 | 18
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 10 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 5
Abdominal Distension (Gastrointestinal disorders) | 4 | 1
Abdominal Pain (Gastrointestinal disorders) | 9 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 8 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 18 | 10
Vomiting (Gastrointestinal disorders) | 12 | 4
Asthenia (General disorders) | 6 | 6
Fatigue (General disorders) | 17 | 11
Oedema Peripheral (General disorders) | 7 | 4
Pain (General disorders) | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 3
Urinary Tract Infection (Infections and infestations) | 6 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 1
Blood Creatinine Increased (Investigations) | 3 | 3
Neutrophil Count Decreased (Investigations) | 4 | 4
Platelet Count Decreased (Investigations) | 2 | 9
Weight Decreased (Investigations) | 3 | 3
White Blood Cell Count Decreased (Investigations) | 6 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Dizziness (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 5
Hypertension (Vascular disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02921919/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT02921919/SAP_001.pdf